CLINICAL TRIAL: NCT04383405
Title: Aquatic Therapy During Post-acute Intensive Neurorehabilitation in Patients With Severe Traumatic Brain Injury: a Preliminary Randomized Controlled Trial
Brief Title: Aquatic Sequential Preparatory Approach and Severe Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, head of rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE/PROG775/2019SPA
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Traumatic Brain Injury; Severe Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential Preparotory Approach (Experimental)
  Interventions: Other: Aquatic Training
- Conventional (Active Comparator)
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Aquatic Training — Aquatic Training training consists of a sequential and a preparatory approach aimed at enhancing dynamic postural stability. The exercises follow a specific sequence starting from a kneeling position, proceeding to a sitting position and ending with a supine position. Step exercises preparatory for gait were performed using a step and two floating aids. Gait exercises were performed first with the upper limbs placed on two floating aids and then during a dual motor task (i.e. catching a ball thrown by the therapist). Subjects performed three sessions a week for four weeks and each session lasting 45 minutes. The training was carried out by a physiotherapist who had at least 5 years of experience in aquatic neurorehabilitation.
  Arms: Sequential Preparotory Approach
Other: Conventional Training — Conventional land-based therapy consists of customized exercises focused on static and dynamic postural stability improvement. The exercises included the active-assisted mobilization, the muscle stretching the postural transition, the balance and the gait training. The control approach was carried out three times a week for four weeks and each session lasted 45 minutes.
  Arms: Conventional

SUMMARY:
Traumatic brain injury (TBI) is an acquired insult to the brain from an external mechanical force. It is considered a major cause of mortality and of long-term disabilities in young adults, especially considering high-income countries.

The TBI can cause a wide range of temporary and/or permanent brain's dysfunctions that can involve physical, cognitive, behavioural and emotional functioning limiting everyday life and social activities and leading to a lowers quality of life.

a sequential preparatory approach (SPA), performed in aquatic environment, based on increasing difficulty and following a specific sequence of preparatory exercises (from the simplest to the most complex) could be an effective complementary training during post-acute intensive rehabilitation in patients with severe traumatic brain injury (sTBI).

ELIGIBILITY:
Inclusion Criteria:

* age between 15 and 65 years;
* Glasgow coma scale (GCS) score ≤ 8 (used to objectively describe the severity of impaired consciousness at the time of injury)
* level of cognitive functioning (LCF) ≥7;
* ability to understand verbal commands.
* acclimatization to water.

Exclusion Criteria:

* Cognitive deficits affecting the ability to understand task instructions (Mini-Mental State Examination > 24);
* Severe unilateral spatial neglect (diagnosed with a test battery that included the Letter Cancellation test, Barrage test, Sentence Reading test and the Wundt-Jastrow Area Illusion Test);
* Severe aphasia (diagnosed by means of neuropsychological assessment);
* Presence of other neurological diseases;
* Presence of cutaneous and mycosis infections;
* Presence of open wounds, eczema, skin ulcers, decubitus lesions, severe burns;
* Presence of PEG (Percutaneous endoscopic gastrostomy);
* Presence of tracheostomy;
* Urinary incontinence;
* Presence of otitis
* Presence of orthopedic or cardiac comorbidities that would limit participation in the experimental and conventional training (all of which were clinically evaluated).

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Berg Balance Scale (BBS) at 1month | 1 month
  Change of Berg Balance Scale (BBS) from baseline at 1 month. BBS values ranging from 0 to 56, where 0 means the lowest level of function and 56 the highest

SECONDARY OUTCOMES:
Tinetti Balance and Gait Scale (TBG) | baseline and after 4 weeks of training
  Change of Tinetti Balance and Gait Scale (TBG) from baseline at 4 weeks of training and at 4 weeks after the end of the training. TBG values ranging from 0 to 28, where 0 means the worse outcome and 28 the best one.
Modified Barthel Index (MBI) | baseline and after 4 weeks of training
  Change of Modified Barthel Index (MBI) from baseline at 4 weeks of training and at 4 weeks after the end of the training. MBI values ranging from 0 to 105, where 0 means the worse outcome and 105 the best one.
Modified Ashworth Scale (MAS) | baseline and after 4 weeks of training
  Change of Modified Ashworth Scale (MAS) from baseline at 4 weeks of the training and at 4 weeks after the end of the training. MAS values ranging from 0 to 5, where 0 means the best outcome and 5 the worse one.
Change in quality of life assessed by the proxy version of the Quality of Life after Brain Injury (Proxy-QOLIBRI) | baseline and after 4 weeks of training
  Change of proxy version of the Quality of Life after Brain Injury (Proxy-QOLIBRI) from baseline at 4 weeks of training and at 4 weeks after the end of the training. (Proxy-QOLIBRI) values ranging from 0 to 100, where 0 means the worse outcome and 100 the best one.
Disability Rating Scale (DRS) | baseline and after 4 weeks of training
  Measure of function after TBI intended to measure function from "coma to community." Minimum score= 0; Maximum score= 29 (High scores are indicative of greater degree of disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tramontano, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided